CLINICAL TRIAL: NCT03694236
Title: Concurrent Neoadjuvant Chemoradiotherapy Plus Durvalumab (MEDI4736) in Resectable Stage III NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0353
Record Dates: First submitted 2018-08-14; First posted 2018-10-03 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Potentially Resectable Stage II/IIIa NSCLC
Keywords: NSCLC; Durvalumab; medi4736
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab (Experimental): This study is single arm phase II study to evaluate efficacy and safety of durvalumab and chemoradiotherapy (paclitaxel and carboplatin) in treatment-naïve clinical stage II/IIIa NSCLC.
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — Neo-adjuvant chemoradiation period The treatment consisted of paclitaxel, carboplatin, duvalumab and radiation. The radiation treatment comprises 45Gy (total 25Fr) and that will be about 5 weeks. Intensity modulated RT (IMRT) or 3D CRT (three-dimensional conformal radiotherapy) will be allowed.
  Surgery Chest CT and/or PET CT with appropriate other diagnostic method (ex. Bronchoscopy) will be performed before surgery and type of surgery Follow-up period There is every 4 month visit with chest CT and abdominal CT is done at 1,2,5 post-op year. Other diagnostic method can be performed if indicated.

SUMMARY:
Combination treatment of Durvalumab with chemoradiotherapy is ongoing for head/neck cancer, renal cell carcinoma, melanoma, and non-small cell lung cancer (NCT02318771) and pancreatic cancer (NCT02305186).Combining Durvalumab with neoadjuvant chemoradiotherapy is a promising strategy to improve clinical outcome in stage III lung cancer. Using serial biopsied and surgically resected fresh tissue through the novel/high-throughput RNA sequencing technologies, we want to identify the change immune signature in tumor microenvironment of NSCLC patients after Durvalumab treatment. With hypothesis that PD-1 inhibitor as a component of neoadjuvant chemoradiotherapy followed by surgery could increase complete pathologic response rate and disease free survival, and overall survival, we suggest adding Durvalumab to neoadjuvant chemoradiation in stage II/III resectable NSCLC. And with immune marker study using FACS, whole exome sequencing, or RNAsequencing, we can find the potential predictive biomarker for anti-PD-L1 blockade. And in this study, we can get "whole" surgical specimen not biopsy sample after Durvalumab treatment so the analysis for immune marker, tumor microenvironment, and various tumor infiltrating immune cells and their changes will be available.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects must fulfill all of the following criteria:

1. Histologically confirmed NSCLC
2. Clinical stage III (including N2 stage and potential candidate for resection)
3. Written informed consent and any locally-required authorization (IRB) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
4. Age > 20 years at time of study entry
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500μL
   * Platelet count ≥ 100,000μL
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). <This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

     * Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

--Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL) 6. Life expectancy of 6 months 8. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥50 years old and no menses for 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Patients with metastatic lesions or clinical N3 lymph nodes
2. Participation in another clinical study with an investigational product during the last 60 months
3. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) Previous enrollment in the present study
4. Any previous treatment (chemotherapy, radiotherapy or surgery) to current disease - NSCLC
5. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
6. History of leptomeningeal carcinomatosis
7. Brain metastases or spinal cord compression. Subjects with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
8. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 36months prior to the first dose of study drug
9. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
10. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
11. Current or prior use of immunosuppressive medication within 14days (use 28 days if combining durvalumab with a novel agent) before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, chemotherapy, CT scan premedication)
12. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
13. History of allogeneic organ transplant
14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Subjects with vitiligo or alopecia
    * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
    * Subjects with celiac disease controlled by diet alone
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
16. History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence

    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
    * Adequately treated thyroid cancer (except. Anaplastic thyroid cancer)
17. History of primary immunodeficiency
18. Active pulmonary tuberculosis (Patients with old tuberculosis can be enrolled) Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
19. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
20. 21. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
21. History of hypersensitivity to the combination or comparator agent
22. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
23. Inability to comply with protocol or study procedures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | for 6 weeks
  To evaluate pathologic complete response (pCR) rate

SECONDARY OUTCOMES:
Objective response rate (ORR) | from date of randomization until the date of first documented progression, assessed up to 5 years
DFS (disease free survival) | from date of randomization until the date of first documented progression, assessed up to 5 years
OS (overall survival) | from date of randomization until the date of first documented progression, assessed up to 5 years
clinical and pathologic down staging rate | from date of randomization until the date of first documented progression, assessed up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided